CLINICAL TRIAL: NCT06953180
Title: Epigenetics and Prevention of Non-communicable Diseases in Kazakhstan: a Personalized Approach and Biological Age Prediction
Brief Title: Epigenetics and NCD Prevention in Kazakhstan: Personalized Approaches and Biological Age Prediction
Status: Recruiting | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Vice-rector, Asfendiyarov Kazakh National Medical University
Other Study IDs: BR27304987
Record Dates: First submitted 2025-03-31; First posted 2025-05-01 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases (CVD); Type 2 Diabetes; Chronic Respiratory Diseases; Obesity (Disorder); Chronic Kidney Diseases
Keywords: DNA methylation; precision medicine; preventive medicine; artificial intelligence; biomedical modeling
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Obesity; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples and peripheral blood mononuclear cells (PBMCs) will be collected. DNA will be extracted and analyzed for telomere length (via quantitative real-time polymerase chain reaction (qPCR)) and methylation patterns (using methylation-sensitive high-resolution melting (MS-HRM)). Only high-quality DNA (assessed by spectrophotometry and fluorometry) will be retained. Samples will be stored at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study includes 1 cohort divided into 4 age subgroups.: The study follows a multistage cluster sampling design with age and gender stratification. A total of 1 cohorts have been identified, further divided into 4 age subgroups:
  1. 18-29 years
  2. 30-44 years
  3. 45-59 years
  4. 60-69 years Each age group is designed to have an equal distribution of men and women, ensuring gender balance across all subgroups.
  Interventions: Other: Genetic: DNA analysis

INTERVENTIONS:
Other: Genetic: DNA analysis — Investigation of telomere length (TL) and DNA methylation level analysis

SUMMARY:
This study aims to enhance personalized and preventive care for non-communicable diseases (NCDs) in Kazakhstan by examining epigenetic factors, predicting biological age and reproductive function using machine learning, and developing health improvement recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 69 years.
* Residents of 17 regions of Kazakhstan.
* Willingness to participate and provide informed consent.

Exclusion Criteria:

* Age less than 18 years old or over 69 years old.
* Failure to provide informed consent or incomplete participation in data collection procedures.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of 6,720 adult volunteers aged 18 to 69 years, residing across 17 regions of Kazakhstan. Participants are stratified by age and gender to ensure balanced representation within the following age groups:
  * 18-29 years
  * 30-44 years
  * 45-59 years
  * 60-69 years Each age group includes an equal proportion of men and women, ensuring gender balance. The selection follows a multistage cluster sampling design, incorporating various socioeconomic backgrounds and health statuses to enhance the generalizability of findings.
Sampling Method: Probability Sample
Enrollment: 6720 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Machine Learning Model for Predicting Biological Age | Within 10 months from start of data collection
  Evaluation of the model's performance (based on telomere length and DNA methylation) using Mean Absolute Error (MAE), Mean Squared Error (MSE), and R².
Accuracy of Reproductive Function Prediction Model | Within 10 months from start of data collection
  Development and validation of machine learning model to predict reproductive function using biomarkers. Model performance evaluated via MAE, MSE, and R².

CONTACTS AND LOCATIONS:
Locations (1):
- Asfendiyarov Kazakh National Medical University, Almaty, Kazakhstan, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided